CLINICAL TRIAL: NCT06489002
Title: DEDICATE: aDvancing carE Management aDoption In Community heAlTh cEnters
Acronym: DEDICATE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OCHIN, Inc. (Other)
Responsible Party: Principal Investigator, Nicole Cook, Principal Investigator, OCHIN, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 00074727
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Social Determinants of Health; Primary Care; Diabetes Mellitus, Type 2; Hypertension
Keywords: Social Determinants of Health; Implementation support; Primary Care; Electronic health records
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension

STUDY DESIGN:
Intervention Model Description: A stepped-wedge cluster randomization design will be used to assess the impact of implementation support strategies to support social needs screening and referrals for patients in care management.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Intervention health centers will receive implementation support when they crossover from Control to Intervention.
  Interventions: Other: Implementation Support
- Control Arm (No Intervention): Control health centers will not receive an intervention prior to crossover to Intervention.

INTERVENTIONS:
Other: Implementation Support — Health centers receiving the intervention will have access to implementation support strategies designed to support adoption of social needs screenings and referrals to community organizations for patients with unmet social needs receiving care management. Implementation support will be provided by an OCHIN trainer, practice facilitators, workflow engineer, and analysts.
  Arms: Intervention Arm

SUMMARY:
DEDICATE will refine and test the effectiveness of evidence-based implementation support strategies designed to support care management teams' sustained use of electronic health record (EHR)-based functionalities to address unmet social needs through improved clinical-community linkages. This study will test the hypothesis that providing implementation support to health center care management teams will lead to increased adoption of EHR functionalities and increased social needs screenings and referrals to community organization to address unmet social needs through a cluster-randomized trial. This study's results will have implications for patients with social needs receiving care management in primary care settings.

DETAILED DESCRIPTION:
The investigators will use a hybrid effectiveness-implementation mixed methods design to assess the impact of evidence-based implementation support strategies designed to support the care management teams' adoption of EHR functionalities that enable social needs screening and referrals to community organizations. After conducting a three-month pilot study with three health centers to test and refine the implementation support strategies, 20 community-based health centers will be recruited to participate in a stepped-wedge, cluster-randomized trial. Eligible OCHIN health centers include those that provide primary care, use an EHR-based care management tool for at least one care management or population health program that addresses social needs for a monthly average of > 15 enrolled patients. Once 20 health centers have been enrolled, health centers will be randomized to one of five wedges for staggered receipt of the intervention. This method will allow us to provide tailored support to four health centers at a time and enables all health centers to eventually receive the intervention. Participating sites will be provided implementation support strategies for using EHR-based functionalities to conduct screening and referrals for patients with social needs. Participating sites will be followed after receiving the intervention until Y4Q4 to assess primary and secondary outcomes.

Implementation strategies to support adoption of EHR-based functionalities for social needs activities by care management teams in health centers comprises the intervention. The intervention will be delivered to health center care management staff outside of patient care. Patients will not directly receive the intervention and will continue to receive regular care from the health center. For all study health centers, quantitative data will be collected (via EHR data extraction) on care team use of EHR functionalities and social risk screening and coordination provided by care teams. Limited clinical data will be collected on patients seen at a study health centers during the study period. Qualitative data will also be collected, including semi-structured interviews with clinic staff from all enrolled study sites.

NOTE: Individual patients will not be assigned to an intervention. Instead, randomization and intervention will occur at the health center level.

ELIGIBILITY:
Inclusion Criteria

• Health centers that use an EHR-based care management tool for at least one care management or population health program that addresses social needs for a monthly average of > 15 enrolled patients

Exclusion Criteria

* Health center participated in pilot
* Health center is a school-based health center
* Health center provides care to prison population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Social needs screening | From six months prior to the intervention, assessed up to 12 months.
  Binary variable of whether the patient has been screened for social needs
Social needs referral | From six months prior to the intervention, assessed up to 12 months.
  Binary variable of whether patients with unmet social needs received referrals to a community organization

SECONDARY OUTCOMES:
Community-based services receipt for referred social needs | From six months prior to the intervention, assessed up to 12 months.
  Binary outcome of receipt of community services (closed-loop referral) among patients with social needs who were referred to community organizations
Controlled hypertension | From six months prior to the intervention, assessed up to 12 months.
  Binary outcome of blood pressure control (defined as <140/90) at the most recent visit among patients with hypertension
Controlled type 2 diabetes mellitus | From six months prior to the intervention, assessed up to 12 months.
  Binary outcome in HbA1c control (defined as <9%) at the most recent visit among patients with diabetes mellitus

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Gold, PhD, Principal Investigator — OCHIN, Inc.; Nicole Cook, PhD, Principal Investigator — OCHIN, Inc.

IPD SHARING:
Plan to Share IPD: No
All EHR data are proprietary to the OCHIN health centers and thus will not be made directly available beyond the study team.

REFERENCES:
- [Derived] Cook N, Gunn R, McGrath BM, Donovan J, Pisciotta M, Owens-Jasey C, Fein HL, Templeton A, Larson Z, Gold R. Implementation strategies to improve adoption of screening and linkages for non-medical drivers of health in care management using enabling technologies: study protocol for a cluster randomised trial. BMJ Open. 2025 Nov 5;15(11):e100340. doi: 10.1136/bmjopen-2025-100340. PMID 41198205
- [Derived] Cook N, Pisciotta M, Larson Z, Fein HL, Donovan J, McGrath BM, Gunn R, Owens-Jasey C, Templeton A, Volk-Britton M, Nishiike Y, Stowe S, Gold R. Using a Modified Delphi Process to Develop an Intervention to Support Care Coordination of Patient Social Needs in Primary Care. J Adv Nurs. 2025 Aug 1:10.1111/jan.70109. doi: 10.1111/jan.70109. Online ahead of print. PMID 40747910
- [Derived] Cook N, Gunn R, McGrath BM, Donovan J, Pisciotta M, Owens-Jasey C, Fein HL, Templeton A, Larson Z, Gold R. Implementation strategies to improve adoption of unmet social needs screening and referrals in care management using enabling technologies: study protocol for a cluster randomized trial. Res Sq [Preprint]. 2024 Oct 17:rs.3.rs-4985627. doi: 10.21203/rs.3.rs-4985627/v1. PMID 39483896